CLINICAL TRIAL: NCT01576315
Title: Efficacy of Itraconazole and of Voriconazole in Patients With Cystic Fibrosis and Presenting With Persistent Positive Sputums for Aspergillus.
Brief Title: ATCF (Azole Therapy in Cystic Fibrosis)
Acronym: ATCF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-005799-41
Record Dates: First submitted 2012-03-29; First posted 2012-04-12 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cystic Fibrosis; Aspergillus Infections
Keywords: cystic fibrosis; Aspergillus; itraconazole; voriconazole
MeSH Terms: conditions — Cystic Fibrosis; Aspergillosis | interventions — Itraconazole; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- itraconazole (Experimental): * itraconazole 10 mg/mL oral solution
  * patients > 40 kg body weight : 200 mg morning and evening.
  * patients < 40 kg body weight : 100 mg morning and evening.
  * dosage out of meal.
  * Without a loading dose
  Interventions: Drug: Itraconazole/voriconazole
- voriconazole (Experimental): * voriconazole 40 mg/mL oral suspension :
  * patients > 40 kg body weight : 200 mg morning and evening.
  * patients < 40 kg body weight : 100 mg morning and evening.
  * dosage out of meal.
  * Without a loading dose
  Interventions: Drug: Itraconazole/voriconazole

INTERVENTIONS:
Drug: Itraconazole/voriconazole — The two treatments will be administered orally for 6 months One doage of treatment permitted based on plasma levels will be performed after two weeks of treatment.
  Other Names: Non applicable.

SUMMARY:
Aspergillus infection is an infectious complication which frequently occurs in cystic fibrosis. The efficacy of azole therapy in patients with cystic fibrosis with persistent positive sputums for Aspergillus is still unknown. Furthermore, the efficacy of itraconazole and voriconazole in this indication has never been evaluated in a large prospective controlled clinical trial, even though many teams already use it. The ATCF study aims to assess in patients with cystic fibrosis with persistent Aspergillus positive cultures the efficacy of itraconazole and voriconazole on the negativisation of the sputum cultures for Aspergillus.

DETAILED DESCRIPTION:
Aspergillus infection is an infectious complication which frequently occurs in cystic fibrosis. The efficacy of azole therapy in patients with cystic fibrosis with persistent positive sputums for Aspergillus is still unknown. Furthermore, the efficacy of itraconazole and voriconazole in this indication has never been evaluated in a large prospective controlled clinical trial, even though many teams already use it.

The ATCF study is a prospective, multicenter, randomized, open-label, controlled phase II trial, performed in patients with cystic fibrosis with persistent Aspergillus positive cultures.

The primary outcome is to assess the efficacy of itraconazole and voriconazole on the course and outcome of the negativisation of the sputum cultures for Aspergillus on two consecutive cultures.

Secondary objectives include the effects of azole therapy on quality of life, FEV1, co-prescription of antibiotic and steroids, plasma concentrations of antifungal agents, speed of negativisation of sputum culture for Aspergillus, outcome of other diagnostic criteria (Aspergillus detection by PCR, precipiting antibodies, total and specific IgE, eosinophilia), and the safety profiles of the two products. Mycological failures, and impact of anti-fungal treatments on lung and systemic inflammation will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cystic fibrosis,
* men or women,
* age equal greater to 12 years,
* presenting with a positive sputum culture for Aspergillus confirmed twice within 6 months before study entry and at initial visit,
* written informed consent.

Exclusion Criteria:

* patients with a contraindication to one of the antifungal agents evaluated,
* pregnant women or nursing mothers,
* absence of an effective method of contraception in women of child-bearing potential,
* patients with signs or symptoms of invasive aspergillosis,
* patients with signs or symptoms of aspergilloma,
* patients with an infection caused by Burkholderia complex Cepacia or to mycobacteria,
* lung transplant patients, registered on a transplantation waiting list or whose registration is imminent,
* patients who received systemic antifungal therapy for more than 5 days within 2 months prior to inclusion,
* patients currently enrolled in another clinical drug trial,
* ongoing treatment with medicinal products contraindicated with itraconazole and voriconazole or with major interactions which reduce azole concentrations,
* patients treated by medication known to prolong QT interval, or with known prolongation of QTc interval > 450 msec in men and > 470 msec in women,
* Inability to follow or to understand the study procedures.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in percentage of patients with a negativisation of sputum cultures in 2 successive samples | Change from baseline in persentage of patients with a negativisation of sputum cultures at 4, 8, 16, 24 weeks after initiation of therapy
  The primary evaluation criterion is the percentage of patients with a negativisation of sputum cultures in 2 successive samples, according to a standardised technique

SECONDARY OUTCOMES:
plasma concentrations of antifungal agents | at 2 weeks after initiation of therapy
  measurement of plasma concentrations of antifungal agents and testing at 4 weeks in case of dose adjustment.
safety of AFs including measurement of hepatic transaminases | at 2 weeks after initiation of therapy
  safety of AFs including measurement of hepatic transaminases
number of courses of steroids and antibiotics recording | at 2 weeks after initiation of therapy
  number of courses of steroids and antibiotics
quality of life | at 4, 8, 16 and 24 weeks after initiation of therapy
  quality of life self-questionnaire scores, dyspnoea scale scores, 6 minute walking test, FEV1 value, and number of courses of steroids and antibiotics
laboratory test indicators | at 4, 8, 16 and 24 weeks after initiation of therapy
  course of different laboratory test indicators (sputum culture and PCR, IgG, total and specific IgE, eosinophilia)
safety profiles of the antifungal agents | at 4, 8, 16 and 24 weeks after initiation of therapy
  safety profiles of the antifungal agents : impact of anti-fungal treatments on lung and systemic inflammation
mycological failures | after 1 month
  analysis of mycological failures (defined as persistence of a positive culture) by a study over time of the course and outcome of fungal biodiversity of isolates (sequential study of chemosensitivity to different antifungal agents and molecular typing)
number of adverse events recording | at 2 weeks after initiation of therapy
  number of adverse events recording

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Gangneux, MD, PhD, Principal Investigator — Service de parasito-mycologie - Rennes University Hospital
Locations (15):
- France (14):
  - CRCM Adulte et Pédiatrie - Hôpital Nord, Amiens
  - CRCM adulte - Centre Robert Debré, Angers
  - Pediatry - Centre Robert Debré, Angers
  - Pediatric penumologic - Groupe hospitalier de Pellegrin, Bordeaux
  - Pneumology pediatric - Hôpital Femme-Mère-Enfants, Bron
  - CRCM - Pediatry - CHI Créteil, Créteil
  - Service de Pneumologie-Immuno-Allergologie / Hôpital Calmette, Lille
  - Hôpital Nord - Pneumology, Marseille
  - Pneumologie Infantile - Hôpital des enfants, Nancy
  - CRCM - Hôpital Sud, Rennes
  - Pneumology - Hôpital Pontchaillou, Rennes
  - CRCM Pédiatrique - Hôpital de Hautepierre, Strasbourg
  - Pédiatrie - Pneumologie, Allergologie - Hôpital des enfants, Toulouse
  - Pneumology - CH Bretagne-Atlantique, Vannes
- Manchester Adult Cystic Fibrosis Centre - University Hospital of South Manchester, Manchester, United Kingdom

REFERENCES:
- [Result] Gangneux JP, Godet C, Denning DW. Allergic diseases and fungal exposome: Prevention is better than cure. Allergy. 2022 Nov;77(11):3182-3184. doi: 10.1111/all.15436. No abstract available. PMID 35822920
- [Result] Guegan H, Prat E, Robert-Gangneux F, Gangneux JP. Azole Resistance in Aspergillus fumigatus: A Five-Year Follow Up Experience in a Tertiary Hospital With a Special Focus on Cystic Fibrosis. Front Cell Infect Microbiol. 2021 Feb 18;10:613774. doi: 10.3389/fcimb.2020.613774. eCollection 2020. PMID 33680981
- [Result] Guegan H, Poirier W, Ravenel K, Dion S, Delabarre A, Desvillechabrol D, Pinson X, Sergent O, Gallais I, Gangneux JP, Giraud S, Gastebois A. Deciphering the Role of PIG1 and DHN-Melanin in Scedosporium apiospermum Conidia. J Fungi (Basel). 2023 Jan 18;9(2):134. doi: 10.3390/jof9020134. PMID 36836250